CLINICAL TRIAL: NCT05604547
Title: Exploring Near Infrared Spectroscopy (NIRS) Technologies for Assessment of Muscle Physiology, Tissue Oxygenation, and Blood Flow in Patients With Sickle Cell Disease (SCD)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000844; 000844-H
Record Dates: First submitted 2022-11-02; First posted 2022-11-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05-13

CONDITIONS: SCD
Keywords: Hemodynamic; Six-Minute Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Single-arm study
  Interventions: Diagnostic Test: Non-Invasive Infrared Spectroscopy

INTERVENTIONS:
Diagnostic Test: Non-Invasive Infrared Spectroscopy — NIRS is a non-Invasive optical technique for characterizing microvascular hemodynamics.

SUMMARY:
Sickle cell disease (SCD) is an inherited disorder of the blood. SCD can injure the smallest blood vessels, which can cause pain and damage organs all over the body. Some treatments are available, but researchers need better ways to monitor the effects of these treatments. An imaging technique called near infrared spectroscopy (NIRS) may be helpful.

Objective:

To test NIRS as a tool for measuring oxygen levels, blood flow, and the makeup of skin and muscle in patients with SCD.

Eligibility:

People aged 18 years and older with SCD. Healthy volunteers are also needed as a comparison for the changes in SCD patients.

Design:

Participants will be screened. They will have a physical exam, and 1 teaspoon of blood will be drawn.

Participants will have NIRS testing on their second visit. Probes will be placed on their skin. A blood pressure cuff will be placed on their arm. The cuff will be filled with air for up to 5 minutes and then released. Participants may be asked to breathe at a certain rate or hold their breath during these measurements.

At this visit, participants will also have an ultrasound exam to get images of their heart. They will be monitored while they walk for 6 minutes. They will have 1 tablespoon of blood drawn. Their height, weight, and vital signs will be measured.

Participants may be asked to return for up to 4 additional visits for NIRS testing within 120 days, but this is optional. The visits must be at least 3 days apart. Each visit will last up to an hour....

DETAILED DESCRIPTION:
Study Description:

This is a non-interventional protocol to explore the role of near infrared spectroscopy (NIRS) technologies as a monitoring tool for assessment of peripheral tissue dynamics in patients with sickle cell disease (SCD). The study will be performed in the outpatient setting. Ethnically-matched healthy subjects will be recruited to participate in baseline NIRS assessments and serve as controls. It is hypothesized that quantitative NIRS will be sensitive to differences in hemodynamic responses between SCD patients and healthy controls in the setting of endothelial dysfunction. In parallel, routine methods of assessing cardiovascular health, including the six-minute walk test, transthoracic echocardiography, and cardiac biomarkers such as pro BNP will be acquired. NIRS holds tremendous potential as a novel point of care test in patients with SCD and may provide further insight on the natural history of the disease and allow for individualized clinical management.

A subset of up to 10 participants in each cohort (SCD patients as well as healthy AA subjects) may be invited to return to the Clinical Center for clinical and NIRS reassessment periodically for a maximum of 4 additional visits, at least 3 days apart, within a 120- day period from their initial (baseline) visit to test repeatability of the NIRS measurements.

Objectives:

Primary Objective:

To quantify baseline hemodynamics in SCD subjects at steady state utilizing NIRS and compare against established clinical/biomarker outcomes, including the six-minute walk test, transthoracic echocardiogram and pro BNP levels.

Secondary Objective:

To compare NIRS measurements in SCD subjects at steady state with NIRS measurements in healthy controls.

Tertiary Objective:

To quantify baseline hemodynamics in ethnically-matched healthy control subjects (HbAA) utilizing NIRS and compare against established clinical/biomarker outcomes, including the six-minute walk test, transthoracic echocardiogram and pro BNP levels.

Endpoints:

Primary Endpoints:

NIRS measurements that characterize tissue composition, tissue metabolism, and blood flow will be collected in SCD subjects in steady state. Primary endpoints include:

* Oxy-/deoxy- hemoglobin concentration for assessing tissue composition
* Tissue oxygen saturation for assessing tissue metabolism
* Blood flow index: Post-occlusion hyperemic response for describing endothelial function.

We will examine correlations between these endpoints and biomarker and clinical endpoints among SCD participants to assess the extent to which NIRS measurements may capture clinical features of SCD.

Secondary Endpoints:

The same endpoints described above will be collected from healthy controls and used to assess differences in tissue composition, tissue metabolism, blood flow between SCD subjects and controls.

Tertiary Endpoints:

To evaluate the tertiary objective of characterizing NIRS responses in healthy controls we will collect:

* Oxy-/deoxy- hemoglobin concentration for assessing tissue composition
* Tissue oxygen saturation for assessing tissue metabolism
* Blood flow index: Post-occlusion hyperemic response for describing endothelial function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Sickle Cell Disease

* Individuals with confirmed sickle cell disease (HbSS and S beta 0 genotypes)
* 18 years of age and older
* Willingness and capacity to provide informed consent
* Individuals must be on stable does of Hydroxyurea for 90 days prior to baseline visit

Ethnically matched controls

* Individuals with HbAA genotype
* 18 years of age and older
* Willingness and capacity to provide informed consent

EXCLUSION CRITERIA:

Sickle Cell Disease

* Pain crisis requiring parenteral treatment within 4 weeks of screening/enrollment
* Blood transfusion within 60 days or exchange transfusion within 90 days of screening/enrollment
* Use of Oxbryta (voxelotor), Adakveo (crizanlizumab), and/or Endari (L-glutamine) within the 12 weeks prior to signing consent
* Women who are currently pregnant
* Presence of an arterial-venous shunt, recent axillary node dissection, or any deformity or surgical history that interferes with proper access for brachial cuff occlusion procedure of the extremities
* Mobility difficulties causing the inability to complete 6-minute walk test

Ethnically matched controls

* Women who are currently pregnant
* Presence of an arterial-venous shunt, recent axillary node dissection, or any deformity or surgical history that interferes with proper access for brachial cuff occlusion procedure of the extremities
* Mobility difficulties causing the inability to complete 6-minute walk test
* Blood transfusion within 60 days or exchange transfusion within 90 days of screening/enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to enroll 20 individuals in each of the following participant groups: SCD (20 HbSS/S-beta0) and 20 healthy controls (genotype HbAA) To obtain this level of enrollment we request a screening ceiling of 60 individuals (30 people per each group) for an enrolment target of 20 SCD and 20 healthy controls who complete participation. Twenty individuals per group should help identify specific hypotheses for testing and estimates of variability and effect size. Correlations between NIRS measurements and clinical/biomarker measurements will need to be relatively strong to meet statistical significance criteria at a 5 percent alpha level for a two-sided test. Assuming data have a bivariate normal distribution, a true correlation of 0.5 and 0.6 are associated with power of 64 percent and 84 percent, respectively. If a Spearman correlation test is used instead of a Pearson correlation (if distribution appear non-normal) then power falls to 58 percent and 76 percent, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
To quantify baseline hemodynamic function in SCD subjects at steady state utilizing NIRS in parallel with clinical assessments of cardiovascular function, including the 6-minute walk test (6MWT), pro BNP levels and transthoracic echocardiogram. | 120 days
  Baseline NIRS measurements will permit real time assessment of peripheral tissue hemodynamics, including oxygenation and blood flow, in relation to established markers of cardiovascular health in subjects with SCD, including the 6MWT, TTE, and pro BNP levels

SECONDARY OUTCOMES:
To assess baseline tissue hemodynamic function utilizing NIRS in ethnically-matched healthy control subjects without (AA) and with sickle cell trait (AS) as compared to baseline NIRS assessments in patients with SCD. | 120 days
  This will permit comparison of peripheral tissue hemodynamics, including blood flow and oxygenation, and cardiovascular clinical outcomes (6MWT, TTE, pro BNP) in subjects with SCD and ethnically-matched healthy volunteer subjects. NIRS results may validate abnormal tissue hemodynamic responses observed in subjects with SCD as compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000844-H.html

DOCUMENTS (1):
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT05604547/ICF_000.pdf